CLINICAL TRIAL: NCT07265323
Title: Effect of Physiologic Insulin Intervention on Insulin Sensitivity and Cognition
Brief Title: Effect of Physiologic Insulin Administration on Insulin Sensitivity and Cognition
Acronym: MIND-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Tim Gilbert, Principal Investigator, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-019-PBRC; PBRC Foundation funds (Other: Pennington Biomedical Research Foundation)
Record Dates: First submitted 2025-11-18; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer s Disease; Alzheimer Blood Biomarkers; Insulin Sensitivity
Keywords: Alzheimer's disease; Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physiologic Insulin (Experimental): Insulin infusion at five-minute intervals over approximately two hours weekly for six months. Initially infusion will be weekly and then frequency will reduce based on participants' response.
  Interventions: Other: Physiological Insulin Intervention

INTERVENTIONS:
Other: Physiological Insulin Intervention — Insulin infusion every five minutes over approximately two hours for six months. Initially infusion will be weekly and then frequency will reduce based on participants' response.

SUMMARY:
The goal of this clinical trial is to determine if a weekly delivery of insulin at short intervals lasting up to 2 hours can improve insulin sensitivity and cognition in adults with Alzheimer's Disease. It will also provide information about the safety and feasibility of this intervention.

The main questions it aims to answer are:

Does the intervention improve insulin sensitivity (how the body uses glucose)?

Does the intervention improve cognition, measured by the Montreal Cognitive Assessment (MoCA) and the Revised Memory and Behavior Problems Checklist (RMBPC)?

What changes occur in brain glucose uptake (FDG-PET)?

Participants will:

Receive the intervention once a week for 6 months, with each session lasting up to 2 hours

Complete cognitive assessments. Adverse events will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Mini Mental State Examination (MMSE) score < 25

Exclusion Criteria:

* On daily medication for the specific treatment of anxiety including benzodiazepines.
* An infant, child, or teenager
* A pregnant woman
* A prisoner
* Having any condition that impedes testing of the study hypothesis or are otherwise deemed to be unsuitable (determined by the investigative team).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Cognition | Over a six-month period
  Cognition will be assessed using Montreal Cognitive Assessment (MoCA). The MoCA test scores range from 0 to 30, with a higher score indicating a better outcome.
Cognition | Over a six-month period
  Cognition will be assessed using the Revised Memory and Behavior Problems Checklist (RMBPC). The two subscales are frequency and reaction. The score for each subscale ranges from 0 to 96. A lower score indicates a better outcome.
Insulin Sensitivity | Over a six-month period
  Insulin sensitivity (glucose disposal rate measured during a hyperinsulinemic euglycemic clamp)

SECONDARY OUTCOMES:
Brain Glucose Uptake | Six months
  We will measure brain glucose uptake using FDG-PET.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Gilbert, M.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No